CLINICAL TRIAL: NCT07152951
Title: Prevalence of Electrolyte Disturbances in Infants and Children With Gastrointestinal Diseases
Brief Title: Electrolytes Disturbance in Infant
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Arwa Hosny Hammam Hasanien, Resident doctor, Assiut University
Other Study IDs: AssuitUniversityAUH
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-04

CONDITIONS: Electrolyte Disturbance in Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence of electrolyte disturbances in infants and children with gastrointestinal diseases

DETAILED DESCRIPTION:
Prevalence of electrolyte disturbances in infants and children with gastrointestinal diseases

ELIGIBILITY:
Inclusion Criteria:

* All patients from one month till 4 years who will be admitted to Gastroenterology unit in (AUCH) and diagnosed with a gastrointestinal disease

Exclusion Criteria:

* 1-Neonates >1 month & those <4 years . 2-Patients with acute or chronic kidney diseases that alter electrolyte balance. 3-Patients with endocrine disorders affecting electrolyte balance (e.g adrenal insufficiency). 4-Use of medications that alter electrolyte balance (e.g diuretics, steroids). 5-Critically ill patients that electrolyte disturbance is due to non-gastrointestinal causes.

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients from one month till 4 years who will be admitted to Gastroenterology unit in (AUCH) and diagnosed with a gastrointestinal disease
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
1-Determine prevalence and types of electrolyte disturbances in infants and children with gastrointestinal diseases | From 1 Jan 2025 to 1 Jan 2026

IPD SHARING:
Plan to Share IPD: No